CLINICAL TRIAL: NCT03211156
Title: A Randomized, Double-Blind, Placebo Controlled, Phase 2 Study to Assess Treatment of Gardnerella Vaginalis Vaginal Colonization With Amoxicillin
Brief Title: Treatment of Gardnerella Vaginalis Vaginal Colonization With Amoxicillin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0073
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2017-06-28

CONDITIONS: Vaginitis Gardnerella
Keywords: Amoxicillin; Gardnerella vaginalis; Vaginal Colonization
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo arm (Placebo Comparator): Placebo 2 capsules PO twice a day for 7 days, n=49
  Interventions: Other: Placebo
- Treatment arm (Experimental): Amoxicillin 2 x 250 mg capsules PO twice a day for 7 days, n=49
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin is an aminopenicillin antibiotic
  Arms: Treatment arm
Other: Placebo — Placebo
  Arms: Placebo arm

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 2 study designed to determine if amoxicillin will eradicate vaginal colonization/infection with Gardnerella vaginalis (GV) when administered to women who are colonized/infected with GV but have no clinical evidence of Bacterial Vaginosis (BV). The study will be conducted at 2 clinics in the United States: University of Alabama at Birmingham and Wake Forest University Health Sciences. Entire study duration is approximately 24 months and subject participation duration is approximately 22 days. Approximately 245 healthy adult females, 18 to 45 years of age will be screened to enroll approximately 98 participants to achieve 82 evaluable participants at the test of cure (ToC) visit. Participants will be enrolled and randomized to one of two groups, either amoxicillin (2 x 250 mg capsules by mouth twice daily for 7 days) or placebo. Women who are enrolled will be asked to return for one further visit, Visit 2 (Day 15 - 21), where a ToC will be completed. For those not enrolled, participation will end at their post screening follow up phone call. Women will be asked to use condoms during their participation. The primary objective is to determine if treatment with amoxicillin eradicates GV in women who are colonized/infected with GV but have no clinical evidence of BV.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 2 study designed to determine if amoxicillin will eradicate vaginal colonization/infection with Gardnerella vaginalis (GV) when administered to women who are colonized/infected with GV but have no clinical evidence of Bacterial Vaginosis (BV). The study will be conducted at 2 clinics in the United States: University of Alabama at Birmingham and Wake Forest University Health Sciences. Entire study duration is approximately 24 months and subject participation duration is approximately 22 days. Approximately 245 healthy adult females, 18 to 45 years of age will be screened to enroll approximately 98 participants to achieve 82 evaluable participants at the test of cure (ToC) visit. Women who consent to screening participation will undergo pelvic examination on entry and vaginal specimens collected for pH, whiff test and wet prep microscopy (Amsel criteria with the exception of evaluation of vaginal discharge), Nugent score, nucleic acid amplification test (NAAT) for trichomonas, quantitative NAAT for GV, and microbiome analysis. At Visit 1 (Enrollment - Day 1), women who tested positive for GV by NAAT, negative for BV by Nugent, and negative for trichomonas by NAAT will be enrolled and randomized to one of two groups, either amoxicillin (2 x 250 mg capsules by mouth twice daily for 7 days) or placebo. Women who are enrolled will be asked to return for one further visit, Visit 2 (Day 15 - 21), where a ToC will be completed (a pelvic exam completed with the same specimens taken as those at baseline with the exception of the trichomonas NAAT). For those not enrolled, participation will end at their post screening follow up phone call. Women will be asked to use condoms during their participation. The primary objective is to determine if treatment with amoxicillin eradicates GV in women who are colonized/infected with GV but have no clinical evidence of BV. The secondary objective is to evaluate the safety and tolerability of amoxicillin compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages 18-45, inclusive.
2. No evidence of vaginitis (yeast, trichomonas, and BV/abnormal vaginal flora) or other vaginal conditions which in the opinion of the investigator could be confounders*.

   *These causes will initially be detected by wet mount microscopy with trichomonas during the screening procedures and later confirmed by NAAT and BV/abnormal vaginal flora confirmed by Nugent scoring (Nugent score of 4-10).
3. Presence of GV detected by NAAT*.

   *Results of NAAT testing will be available prior to return for Enrollment visit.
4. Willing to use condoms during vaginal intercourse while participating in the study.
5. Not currently menstruating at screening visit.
6. Willing and able to provide written informed consent.
7. Negative urine pregnancy test on all participants of childbearing potential at study screening.
8. Participant must be of non-childbearing potential* or must be using highly effective birth control** to avoid becoming pregnant.

   *Non-childbearing potential is defined as being post-menopausal for at least 1 year, status after bilateral tubal ligation, or status after bilateral oophorectomy or status after hysterectomy.

   **In addition to the required use of condoms by the male partner during study participation, participants must agree to avoid becoming pregnant by using one of the following acceptable method of birth control for 30 days prior to screening and for the duration of the study:
   * Intrauterine contraceptive device; OR
   * Oral contraceptives; OR
   * Hormonal injections; OR
   * Hormonal implants; OR
   * Contraceptive patches; OR
   * Monogamous relationship with vasectomized partner; OR
   * Exclusively same-sex relationships; OR
   * Abstinence
9. Participant is not planning on taking antibiotics or using any intravaginal microbicides from the Screening visit through the Visit 2 Follow-up (TOC).
10. Participant is willing and able to cooperate to the extent and degree required by this protocol at the discretion of the investigator.

Exclusion Criteria:

1. Pregnant or nursing.
2. Allergic to penicillin, amoxicillin, cephalosporins, or other ß-lactam antibiotic.
3. Use of antibiotics in the past 14 days prior to screening visit.
4. HIV infected.
5. Women taking immunosuppressive agents.

7. History of renal impairment. 8. Use of any investigational drug within the past 30 days prior to screening. 9. Any other condition that, in the opinion of the investigator, would interfere with participation in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - Guilford County Health Department - Greensboro - STD Clinic, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from women who were colonized/infected with Gardnerella vaginalis but have no clinical evidence of Bacterial Vaginosis. Enrollment occurred between 21SEP2017 and 08AUG2019.
Groups:
- Placebo: Participants received Amoxicillin placebo 2 capsules orally twice a day for 7 days, n=49
  Placebo: Placebo
- Amoxicillin: Participants received Amoxicillin 2 x 250 mg capsules orally twice a day for 7 days, n=48
  Amoxicillin: Amoxicillin is an aminopenicillin antibiotic
Period: Overall Study
Arm/Group | Placebo | Amoxicillin
Started | 49 | 48
Received Study Drug | 47 | 45
Completed | 47 | 45
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects, receiving or not receiving the study product, are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Amoxicillin | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (7.8) | 29.0 (7.3) | 29.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 97
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 46 | 44 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 29 | 62
  White | 15 | 13 | 28
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants With Eradication of Gardnerella Vaginalis (GV) in Each Study Arm at Visit 2 (Day 15-21) as Assessed by Nucleic Acid Amplification Test (NAAT).
Description: Eradication of GV is defined by a negative NAAT result for GV at Visit 2. Participants who have a missing GV NAAT result at the test of cure (TOC) visit were classified as treatment failures. The denominator for proportions is based on the number of subjects who were randomized to the specified treatment group.
Time Frame: Day 15 to 21
Population: Participants included in the ITT population are those who randomized, regardless of whether they received study treatment or were compliant with the administration procedures or schedule.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Amoxicillin
Number analyzed (Participants) | 49 | 48
proportion of participants | 0.16 [0.09 to 0.29] | 0.21 [0.12 to 0.34]
Statistical Analysis 1: Comparison: Placebo vs Amoxicillin; Test type: Other; p = 0.757, Chi-squared, Corrected

2. Secondary Outcome: The Proportion of Participants Reporting Related Adverse Events (AEs and SAEs) in Each Study Arm Following the First Dose of Study Product Through Visit 2.
Description: AEs were defined as any untoward medical occurrence in a participant administered a pharmaceutical product. SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. AEs and SAEs were collected from participants following the first dose of treatment through Visit 2 (Day 15-21). Events are included if deemed by the investigator to be related to the study product.
Time Frame: Day 1 through Day 15 to 21
Population: Participants included in the safety population are those who randomized and received at least one dose of treatment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Amoxicillin
Number analyzed (Participants) | 47 | 45
proportion of participants | 0.04 [0.01 to 0.14] | 0.18 [0.08 to 0.32]
Statistical Analysis 1: Comparison: Placebo vs Amoxicillin; Test type: Other; p = 0.048, Fisher Exact

ADVERSE EVENTS:
Time Frame: Unsolicited non-serious AEs and SAE were collected through Visit 2 (Day 15-21) after the first dose of treatment.
Description: The safety data collection was targeted to collect serious and non-serious adverse events and congenital anomalies / birth defects as applicable that occurred after the first dose of treatment through Visit 2 (Day 15-21). Adverse events were captured by subject report/interview and clinical assessments, including clinician-conducted pelvic examination.
Arm/Group | Placebo | Amoxicillin
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/45
Other Adverse Events (participants affected / at risk) | 3/47 | 10/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Amoxicillin (N=45)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Allergic reaction to excipient (Immune system disorders) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 2 (2)
Potassium hydroxide preparation positive (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03211156/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03211156/SAP_001.pdf